CLINICAL TRIAL: NCT04837417
Title: Deficit in Quadriceps Voluntary Activation After Anterior Cruciate Ligament Reconstruction: Roles of the "Learned Non-use" Paradigm and the Interhemispheric Inhibition
Acronym: AQUARIUS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: ASST Gaetano Pini-CTO (Other)
Responsible Party: Sponsor
Other Study IDs: 24C021_2020
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Anterior cruciate ligament reconstruction; acquired non-use; voluntary activation; quadriceps femoris; rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pathologic group: At least 10 male participants who underwent anterior cruciate ligament arthroscopic reconstruction using semitendinosus and gracilis tendons graft, between 6 and 18 months before the tests
  Interventions: Diagnostic Test: Pathologic group

INTERVENTIONS:
Diagnostic Test: Pathologic group — Voluntary Activation level will be determined with the interpolate twitch technique (ITT), both during isometric contractions (knee at 40° flexion) and during isokinetic contraction at angular velocity equal to 100°/s.
  Vastus Medialis and Soleous H-reflex will be measured. Cortical excitability and interhemispheric connectivity will be measured through transcranial magnetic stimulation (TMS).
  Tests of balance in standing will be performed using the EquiTest platform. Individuals will be requested to perform three different tasks: Sensory Organization test, Adaptation Test upward/downward, Motor Control test backward/forward. Surface electromyography from lower limbs will be recorded.
  Through TMS driven by neuronavigation, the cortical representation of the Quadriceps muscle will be studied.
  Gait analysis will be performed on a treadmill mounted on force sensors. Participants will walk at increasing velocities from 0.4 m/s to 1.6 m/s. Speed will be increased of 0.2 m/s every 30 s.

SUMMARY:
Anterior cruciate ligament (ACL) tear is mainly caused by sport injuries. 40% of injuries are attributed to noncontact mechanisms involving pivoting. Regaining quadriceps strength is a primary focus of patients pursuing a rehabilitation program after ACL reconstruction (ACLR). Unfortunately, despite rehabilitation programs aimed at reversing this muscle weakness, quadriceps strength deficits may persist for years. Moreover, this deficit leads to increased risk of sustaining another knee injury, and increased risk for developing posttraumatic osteoarthritis. At present, neither the optimal rehabilitative program nor the clinical and instrumental parameters to take into account at the time of return to activity have reached a consensus among clinicians.

The investigators hypothesize that:

* a persistent deficit in voluntary activation, that is an inability to achieve complete activation of a muscle, is present after ACLR.
* this deficit in voluntary activation is associated with a phenomenon of "learned/acquired non-use" both in balance and during gait. This phenomenon will be demonstrated by investigating asymmetries in the recruitment of the injured lower limb in balance tests and during gait.
* the "learned/acquired non-use" paradigm is associated to asymmetries in the hemispheric cortical activity. This phenomenon will be investigated through transcranial magnetic stimulation.

The primary endpoint is the demonstration that the quadriceps muscle weakness after ACLR may represent a case of "learned non-use". This behaviour looks automatic and unconscious, so that the adjective "acquired" seems preferable to "learned". It consists of the under recruitment of the impaired side, once healed, as a form of unconscious protection, which is adopted when the contralateral side may carry out the function.

The secondary outcome is the investigation of the correlation among the deficits in voluntary activation, in balance tests, during gait, and in the neurophysiologic trials, with the clinical conditions of the patients.

It is expected that the injured lower limb show a deficit in the activation of the quadriceps muscle with respect to the contralateral one and with respect to normative data. The impaired limb will present lower recruitment in balance tests and a deficit in power production during gait.

The contralesional hemisphere will demonstrate higher interhemispheric inhibition, lower short-interval intracortical inhibition (SICI) and higher short-interval intracortical facilitation (SICF) with respect to the ipsilesional hemisphere.

The evidence for an asymmetry between the two lower limbs would support the hypothesis that the "acquired non-use" paradigm has a role in the deficits following ACL lesions and that it is unspecific across asymmetric impairments, and independent of the underlying disease.

Results from the present study will allow:

* the identification of clinical and instrumental criteria to guide the return-to-sport decision following ACLR.
* the estimate of the sample size for future experimental protocols and new rehabilitative programs.

ELIGIBILITY:
Inclusion Criteria:

* anterior cruciate ligament tear with arthroscopic reconstruction, between 6 and 18 months before the tests;
* Tegner activity level > 5;
* Body Mass Index between 18 and 25;
* voluntary knee extension of at least 70°;
* ability to understand the instructions;
* ability to wittingly sign the informed consent form.

Exclusion Criteria:

* other previous knee injuries or surgical interventions;
* major procedures associated with the anterior cruciate ligament reconstruction: osteotomy, other ligaments reconstruction;
* meniscectomy, with surgical removal of more than 30% of the meniscal volume or removal of the meniscal root;
* comorbidities, such as: rheumatic diseases; other congenital or acquired neuromuscular pathologies; diabetes mellitus; osteoporosis; cancer; heart disease; history of epilepsy, endocranial hypertension;
* first degree relatives affected by epilepsy;
* current treatment with oral anticoagulant or antiplatelet therapy;
* drug therapy, which could induce epileptic crisis;
* history of high alcohol consumption;
* implanted electro-sensitive devices;
* implanted intracranial or intraocular metallic devices;
* history of retinal detachment;
* presence of cochlear implant.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The participants will be recruited by ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Presidio Ospedaliero Gaetano Pini, among those who underwent the surgical interventions in the Centre.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Voluntary Activation | Day 1
  Voluntary Activation = [1 - (Interpolated Twitch/Resting Twitch)] percent, where Interpolated Twitch and Resting Twitch are the peak torques caused by the electric shock during the voluntary contraction and at rest, respectively.

SECONDARY OUTCOMES:
H-reflex minimal latency | Day 1
  H-reflex latency is defined as the time it takes for the H-reflex to appear on the EMG relative to the introduction of the stimulus. H-reflex minimal latency represents the minimal latency among the H-reflex amplitudes recorded at the different stimulus intensities.
H/M ratio | Day 1
  H/M ratio is the ratio between H-reflex amplitude and M-wave amplitude.
iSP (Ipsilateral Silent Period) durations | Day 1
  Eight stimuli are applied over the hotspot at an intensity of 140 percent of the stimulator output while subjects are performing a voluntary maximal contraction of the ipsilateral hand, with a figure-of-eight coil for transcranial magnetic stimulation (TMS). Both hemispheres are tested.
  ISP durations are determined by rectifying the EMG traces and averaging them among the 8 stimuli. Baseline EMG is defined as the average value of EMG in the 100 ms before the TMS stimulus. ISP onset is defined as the latency at which the averaged EMG activity became constantly (for at least 10 ms) smaller than the average baseline EMG. ISP offset is set at the first point after ISP onset at which the EMG activity regained the baseline activity for at least 10 ms. ISP duration is defined as: ISPduration = ISPoffset - ISPonset.
iSP (Ipsilateral Silent Period) area | Day 1
  Eight stimuli are applied over the hotspot at an intensity of 140 percent of the stimulator output while subjects are performing a voluntary maximal contraction of the ipsilateral hand, with a figure-of-eight coil for transcranial magnetic stimulation (TMS). Both hemispheres are tested.
  ISParea is computed as the product between baseline EMG and iSP duration.
SICI (Short interval IntraCortical Inhibition) | Day 1
  A paired pulse will be applied over the hand area of the motor cortex to evoke EMG responses in the contralateral muscle. The conditioning stimuli will be given at an intensity of 75 percent of the resting Motor Threshold (rMT) and the test stimuli will be given at an intensity of 120 percent of the rMT. The interstimulus intervals will be 3 and 5 ms. For each interstimulus interval, 8 stimuli will be applied in a random order.
SICF (Short interval IntraCortical Facilitation) | Day 1
  A paired pulse will be applied over the hand area of the motor cortex to evoke EMG responses in the contralateral muscle. The conditioning stimuli will be given at an intensity of 75 percent of the resting Motor Threshold (rMT) and the test stimuli will be given at an intensity of 120 percent of the rMT. The interstimulus intervals will be 15 and 20 ms. For each interstimulus interval, 8 stimuli will be applied in a random order.
SOT score | Day 1
  The patient's task is to maintain an upright stance during 3 20 s trials under six different conditions, including platform and visual surround 'tuned' with individual's sagittal oscillation. The SOT score will be calculated by comparing the sagittal oscillation of the body's centre of mass (COM) to the maximal sagittal oscillation. Score is averaged across the six conditions (range 0 - 100 the higher the score, the lower the oscillation, in each condition).
Map area of quadriceps muscle | Day 1
  Transcranial magnetic stimulation (TMS) will be used to map cortical representation of quadriceps muscle. An optoelectronic neuronavigation system will be used to digitize the scalp stimulation coordinates, to guide the TMS coil to focus on a stimulation site, and to ensure spatial precision during the procedure. Two or three TMS stimuli will be delivered at each of the stimulated scalp sites. The largest peak-to-peak MEP amplitude (mean of three MEPs) across the positions making up the motor map was measured. The map area was defined as the number of scalp positions associated with the mean MEP amplitude larger than 100 μV.
Ankle joint power | Day 1
  Joint kinematics will be recorded through an optoelectronic method as per the Davis anthropometric model. The 3D displacement of the markers will be captured using 10 near-infrared stroboscopic cameras. Joint power will be computed through the spatiotemporal synchronization of ground reaction force vectors and the joint centers of rotation. Only the sagittal plane will be considered for the analysis. Joint power will be computed as the product of joint torque and joint rotation speed. Power will be defined as positive or generated when the joint moment and rotation speed shared the same directions (i. e., when agonist muscles are contracting while shortening), as negative or absorbed otherwise. Positive work will be computed as the integral of the generated (positive) power over time.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Tesio, MD, Full professor, Principal Investigator — Istituto Auxologico Italiano
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano, Milan, MI
  - ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Presidio Ospedaliero Gaetano Pini, Milan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Scarano S, Caronni A, Menon A, Rota V, Amadei M, Perucca L, Brevi E, Maione A, Ferrua P, Tesio L, Randelli PS. Anterior cruciate ligament reconstruction is associated with increased corticospinal excitability and rate of force development. BMC Sports Sci Med Rehabil. 2026 Feb 9. doi: 10.1186/s13102-026-01577-0. Online ahead of print. PMID 41656237